CLINICAL TRIAL: NCT01256996
Title: A Randomized Multicenter Study in the Therapy of Periimplantitis: Scaling Versus Low Abrasive Powder
Brief Title: Therapy of Peri-implantitis: Scaling Versus Low Abrasive Powder
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Heidelberg University (Other)
Responsible Party: Clovis Mariano Faggion Jr. and Marc Schmitter, University of Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MV-329/2009
Record Dates: First submitted 2010-12-02; First posted 2010-12-09 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-10

CONDITIONS: Peri-implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- Low-abrasive powder (Experimental)
  Interventions: Procedure: Air abrasion of the implant surface with a low abrasive powder

INTERVENTIONS:
Procedure: Air abrasion of the implant surface with a low abrasive powder — Test treatment will be performed using the low abrasive powder in a standard air-polishing unit, which will be set up according to the manufacturer's instructions. The unit will be set to a medium water and powder setting, and the powder chamber will be filled to the indicated maximum powder level before treatment to ensure reproducible treatment conditions. The jet will be directed to the periodontal pocket for 5 s per surface (vestibular, lingual, mesio and distal) for subgingival plaque removal.

SUMMARY:
In the last decade, the number of dental implantations continuously increases. However, at the same time, the prevalence of peri-implantitis increases, too. Although both surgical and non-surgical interventions are available for the therapy, there is no efficient and satisfying therapy option resulting in an adequate improvement of this disease.

An innovative, low abrasive powder has been introduced for the therapy of periodontitis. However, the powder might be suitable for the peri-implantitis therapy, also, and could improve the effectiveness of the therapy. The usage of this powder in peri-implantitis patients has not been assessed in a clinical trial although the effectiveness in natural teeth has been demonstrated.

The aim of this prospective, randomised, multi-centre trial is to assess the effectiveness of the aforementioned powder in peri-implantitis patients.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate peri-implantitis
* age ≥18 years
* capacity to contract
* no subgingival debridement within the last six months
* informed consent

Exclusion Criteria:

* pregnancy
* subgingival debridement within the last six months
* bleeding tendency
* usage of antibiotics within the last three months
* insufficient restorations (including caries etc.)
* Diabetes mellitus
* smoker
* implantats with platform switch

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-04 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Pocket probing depth | Twelve months

SECONDARY OUTCOMES:
Assessment of pain levels | One week and six months
Assessment of the oral health related quality of life using the OHIP (14) | One , three, six and twelve months